CLINICAL TRIAL: NCT05548452
Title: Intestinal Microbiota Transplant in Alcohol-Associated Chronic Liver Disease and Cirrhosis: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Intestinal Microbiota Transplant in Alcohol-Associated Liver Disease
Acronym: IMPACT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM20025442; R01AA029398 (NIH)
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Liver Disease; Alcohol-Related; Cirrhosis; Alcohol Use Disorder
Keywords: Intestinal Microbiota Transplant; Alcohol Use Disorder; Cirrhosis; Chronic Liver Disease
MeSH Terms: conditions — Liver Diseases; Fibrosis; Alcoholism | interventions — Fecal Microbiota Transplantation; Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intestinal Microbiota Transplant capsules (Experimental): Capsules will be provided twice during the trial
  Interventions: Drug: Intestinal Microbiota Transplant (IMT) Capsules
- Placebo capsules (Placebo Comparator): Capsules will be provided twice during the trial
  Interventions: Drug: Placebo Capsules

INTERVENTIONS:
Drug: Intestinal Microbiota Transplant (IMT) Capsules — Capsules containing freeze-dried intestinal microbiota from healthy human donors
  Arms: Intestinal Microbiota Transplant capsules
Drug: Placebo Capsules — Capsules containing an inactive substance ("sugar pill")
  Arms: Placebo capsules

SUMMARY:
The purpose of this research study is to test the safety, tolerability, and effectiveness of the capsules that contain bacteria from healthy individuals when used to treat alcohol craving and drinking.

DETAILED DESCRIPTION:
These intestinal microbiota transplant (IMT) capsules are an investigational drug, which means it has not been approved by the U. S. Food and Drug Administration (FDA). In this study, drug name will be compared to placebo (a look-alike inactive substance, a "sugar pill").

Participants will be randomly assigned (like the flip of a coin) to receive either IMT capsules or placebo capsules. Participants have an equal chance of being assigned to any one of the groups.

In this study, participants will be asked to do the following things:

1. Visit VCU medical center up to 8 times for study visits
2. Take either IMT capsule or the placebo, depending upon which group they are assigned to; these capsules will be given twice on enrollment and after one month
3. Have blood drawn, urine and stool collected at each visit
4. Have testing done to determine the speed of brain function
5. Keep a diary at home
6. Take surveys and answer questions about general health, alcohol craving and consumption and how they are feeling.
7. Give permission for the researchers to collect information about liver disease, alcohol and mental health from medical records.

Participation in this study will last up to 7 months.

ELIGIBILITY:
Inclusion Criteria:

->18 years of age

* Advanced liver disease
* Able to give written, informed consent
* Alcohol as a cause of advanced liver disease
* Continued sustained drinking
* Having previously declined a referral to traditional AUD therapy services or having failed such treatments

Exclusion Criteria:

* Lack of sustained drinking
* Recent or current alcoholic hepatitis
* Alcohol withdrawal symptoms
* Clinically significant use of illicit drugs
* Uncontrolled mood disorders or primary psychotic conditions
* MELD score>17
* Unclear diagnosis of chronic liver disease
* Current hepatic encephalopathy on lactulose and/or rifaximin
* WBC count<1000
* Non-elective hospitalization within last month
* on dialysis
* known untreated, in-situ luminal GI cancers
* chronic intrinsic GI diseases (ulcerative colitis, Crohn's disease or microscopic colitis, eosinophilic gastroenteritis and celiac disease)
* Dysphagia within 2 weeks
* History of aspiration, gastroparesis, intestinal obstruction
* Ongoing absorbable antibiotic use
* Severe anaphylactic food allergy
* allergy to ingredients Generally Recognized As Safe in the G3 capsules (glycerol, sodium chloride, hypromellose, gellan gum, titanium dioxide, theobroma oil)
* Adverse event attributable to prior IMT
* ASA Class IV or V
* Pregnant or nursing patients
* acute illness or fever on the day of planned FMT
* Immunosuppression
* Other conditions which make patients are poor candidate for this study per investigator judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of abstinent days | Baseline to 3 months after treatment (analysis of all 3 primary outcomes via Win Ratio)
  Number of drinks per day will be measured through self report
Reduction in WHO drinking levels by 1 or greater at month 3 | Baseline to 3 months after treatment (analysis of all 3 primary outcomes via Win Ratio)
  WHO grade by self report
Phosphatidyl Ethanol (PEth) level change | Baseline to 3 months after treatment (analysis of all 3 primary outcomes via Win Ratio)
  Change to <70

SECONDARY OUTCOMES:
Change in markers of alcohol in urine | Baseline to 3 months after treatment
  Urine samples will be analyzed for levels of Ethyl Glucuronide (EtG) and Ethyl Sulfate (EtS)
Change in markers of alcohol in blood | Baseline to 3 months after treatment
  Blood samples will be analyzed for Phosphatidyl Ethanol (PEth)
Change in percentage of heavy drinking days | Baseline to 3 months after treatment
  Self reported drinking behavior will be used to calculate percentage of heavy drinking days
Change in alcohol craving | Baseline to 3 months after treatment
  The Alcohol Craving Questionnaire is a 12-item instrument
Change in life problems | Baseline to 3 months after treatment
  The Short Index of Problems is a 15-item instrument which measures medical, psychological, social, occupational, and legal problems.
Number of hospitalizations | 6 months
  All hospitalizations and liver-related hospitalizations will be tracked
Number of serious adverse events | 6 months
  All serious adverse events and intervention related adverse events will be tracked
Change in microbial composition | Baseline to 3 months after treatment
  Percentage of beneficial intestinal bacteria will be assessed by genetic analysis of stool samples.
Change in liver function | Baseline to 3 months after treatment
  The Model for end-stage liver disease (MELD) score will be used to asses changes in liver function.
Change in Psychometric hepatic encephalopathy score (PHES) | Baseline to 3 months after treatment
  Brain function will be assessed using the PHES
Change in EncephalApp Stroop Test | Baseline to 3 months after treatment
  Brain function will be assessed using the EncephalApp Stroop Test
Change in health related quality of live (HRQOL) | Baseline to 3 months after treatment
  HRQOL will be assessed using the Sickness Impact Profile

CONTACTS AND LOCATIONS:
Overall Officials: Jasmohan S Bajaj, MD, Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data via NIAAA DA website
Supporting Information: Study Protocol, SAP, ICF